CLINICAL TRIAL: NCT04372225
Title: Predicting Risk Factors of Postoperative Hypocalcemia After Total Thyroidectomy: is Safe Discharge Without Supplementation Possible?
Brief Title: Predicting Risk Factors of Postoperative Hypocalcemia After Total Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Aix Marseille Université (Other)
Responsible Party: Principal Investigator, Paladino Nunzia Cinzia, Principal Investigator, Aix Marseille Université
Other Study IDs: ArixMU
Record Dates: First submitted 2020-04-25; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Hypoparathyroidism
Keywords: thyroidectomy; hypocalcemia; hypoparathyroidism; discharge; PTH
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 477 patients: the biological tests of 477 patients undergoing total thyroidectomy were analyzed
  Interventions: Other: analysis of hypocalcemia

INTERVENTIONS:
Other: analysis of hypocalcemia — analysis of postoperative calcium and PTH levels

SUMMARY:
With increasing economic pressures to shorten the length of hospital stay, there has been much recent interest in studying risk factors for the development of postoperative hypocalcemia.

The aim of this study was to investigate in patients undergoing total thyroidectomy whether serum calcium and/or PTH levels can predict hypoparathyroidism.

DETAILED DESCRIPTION:
Our study consists of analyzing the calcium (mmol/l) and PTH (pmol/l) levels on the first postoperative day. Postoperative treatment with calcium and vitamin D and the length of hospital stay is also taken into consideration.

We also analyze post-operative complications.

ELIGIBILITY:
Inclusion Criteria:

• Total thyroidectomy

Exclusion Criteria:

* concomitant parathyroidectomy for primary hyperparathyroidism
* lobectomy only
* completion thyroidectomy
* central and lateral neck dissection
* patients with calcium and/or vitamin D supplementation prior surgery
* patients with known and significant osteoporosis and renal failure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Analysis of calcium and PTH levels in postoperative day 1
Sampling Method: Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
calcium and PTH thresholds | one years
  For all 477 patients postoperative calcium and PTH levels and treatment with calcium and vitamin D will be analyzed.
  Objective is to identify the calcium and PTH thresholds at which the patient after total thyroidectomy can be discharged without risk of hypocalcemia.

CONTACTS AND LOCATIONS:
Locations (1):
- Conception Hospital, Marseille, France

IPD SHARING:
Plan to Share IPD: No
the data are confidential

REFERENCES:
- [Derived] Paladino NC, Guerin C, Graziani J, Morange I, Loundou A, Taieb D, Sebag F. Predicting risk factors of postoperative hypocalcemia after total thyroidectomy: is safe discharge without supplementation possible? A large cohort study. Langenbecks Arch Surg. 2021 Nov;406(7):2425-2431. doi: 10.1007/s00423-021-02237-2. Epub 2021 Aug 10. PMID 34374848